CLINICAL TRIAL: NCT04966975
Title: Effect and Prognosis of Immunohistochemical Biomarkers Changes in Patients With Bladder Cancer After Neoadjuvant Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Shantou Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SysMU-diag2
Record Dates: First submitted 2021-07-09; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; neoadjuvant chemotherapy; immunohistochemical biomarkers
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Histologically confirmed bladder cancer treated with NAC
  Interventions: Other: neoadjuvant chemotherapy

INTERVENTIONS:
Other: neoadjuvant chemotherapy — The patients receive neoadjuvant chemotherapy for 2-4 cycles before surgery.

SUMMARY:
Clinical trial to investigate the relationship between the expression of immunohistochemical biomarkers GATA-3, CK20, P53 and Ki67 in bladder cancer and pathological complete response after neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
This is a retrospective study included bladder cancer patients treated with neoadjuvant chemotherapy. We analyzed the changes in the expression of GATA-3, CK20, P53 and Ki67 before and after NAC. Evaluating the sensitivity factor for predicting pathological complete response.

ELIGIBILITY:
Inclusion Criteria:

1. Any male or female patient aged 18 or older.
2. Histologically confirmed bladder cancer, cystectomy was performed after NAC.
3. Complete clinical data.

Exclusion Criteria:

1. Patients with severe organic disease who can not tolerate chemotherapy or surgery
2. Patients received previous treatment (chemotherapy, radiation, or molecular targeted therapy).
3. Patients with distant metastasis or other cancer history.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who histologically confirmed bladder cancer treated with neoadjuvant chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Expression of immunohistochemical biomarkers GATA-3, CK20, P53 and Ki67 | 1 year
Tumor regression grade | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jian Huang, MD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No